CLINICAL TRIAL: NCT05229068
Title: A Phase IIIB, Open Label, Non-randomized, Controlled, Multi-country Study to Evaluate Safety, Reactogenicity and Immunogenicity of the Repeat Vaccination With 120 µg Dose of RSV Maternal Vaccine During Subsequent Pregnancy in Healthy Maternal Participants 18-49 Years of Age
Brief Title: A Study of Safety, Reactogenicity and Immune Response of the Repeat Vaccination Against RSV When Given to Female Participants of 18-49 Years of Age During Their Subsequent Uncomplicated Pregnancy
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Following a recommendation from the Independent Data Monitoring Committee of NCT04605159 (RSV MAT 009), GSK made the decision to stop enrolment and vaccination in this study.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 214753; 2021-004012-25 (EudraCT Number)
Record Dates: First submitted 2022-01-27; First posted 2022-02-08 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: Respiratory Syncytial Virus Maternal vaccine; Safety; Reactogenicity; Immunogenicity; Healthy pregnant women; Subsequent pregnancy
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prior_RSV MAT Group (Experimental): Maternal participants who received a single 120 µg dose of RSV MAT vaccine at Day 1 in RSV MAT-004 (NCT04126213), RSV MAT-009 (NCT04605159) or RSV MAT-012 (NCT04980391) parent studies, will receive a single dose of RSV MAT vaccine at Day 1 in the current study and are followed-up until the study end (Day 181 post-delivery).
  Interventions: Biological: RSV MAT
- Prior_Placebo Group (Experimental): Maternal participants who received a single dose of placebo at Day 1 in RSV MAT-004 (NCT04126213), RSV MAT-009 (NCT04605159) or RSV MAT-012 (NCT04980391) parent studies or who did not participate in the parent studies and did not receive any RSV vaccine in the past*, will receive a single dose of RSV MAT vaccine at Day 1 in the current study and are followed-up until the study end (Day 181 post-delivery). *The unvaccinated participants are enrolled if the study cannot enroll sufficient numbers of the maternal participants who received placebo in the parent studies.
  Interventions: Biological: RSV MAT

INTERVENTIONS:
Biological: RSV MAT — Single 120 µg dose of the RSV MAT vaccine reconstituted with NaCl solution, administered intramuscularly in the non-dominant arm, at Day 1.

SUMMARY:
The purpose of this study is to evaluate the safety, reactogenicity and immunogenicity of a single intramuscular dose of the investigational respiratory syncytial virus (RSV) maternal (RSV MAT) vaccine during subsequent uncomplicated pregnancy in maternal participants, 18 to 49 years of age (YOA), who have previously received the RSV MAT vaccine or placebo in the RSV MAT-004 (NCT04126213), RSV MAT-009 (NCT04605159) and RSV MAT-012 (NCT04980391) primary studies.

ELIGIBILITY:
Inclusion Criteria:

Maternal participants

* Only those pregnant participants who received a single 120 µg dose of RSV MAT vaccine or placebo in the RSV MAT-004, RSV MAT-009 or RSV MAT-012 studies OR healthy pregnant participants who had at least one prior live birth and have not received any RSV vaccine in the past.
* Participants who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* Written or witnessed/thumb printed informed consent obtained from the participants prior to performance of any study-specific procedure. The informed consent given at screening should (consistent with local regulations/guidelines) either:

  * include consent for both the maternal participant's participation and participation of the infant after the infant's birth, or
  * include consent for the maternal participant's participation and expressed willingness to consider permitting the infant to take part after the infant's birth (if local regulations/guidelines require parent(s) to provide an additional informed consent after the infant's birth).
  * Both mother and father should consent if local regulations/guidelines require it.
* In good general maternal health as established by medical history and clinical examination before entering into the study.
* Participants between and including 18 and 49 YOA, inclusive at the time of consent.
* Pre-pregnancy body mass index (based on participant's report) 17 to 39.9 kg/m^2, inclusive.
* Singleton pregnancy (including instances where the singleton pregnancy derives from a vanishing twin syndrome).
* Pregnant females at 24^0/7 to 36^0/7 weeks of gestation at the time of study intervention administration (Visit 1), as established by:

  * last menstrual period (LMP) date corroborated by first or second trimester ultrasound examination (U/S) i.e. at or before 28 weeks of gestation.
  * First or second trimester U/S only, if LMP is unknown/uncertain.
  * Certain LMP, corroborated by a U/S performed after 28 weeks of gestation is also acceptable.

NOTE: If pregnancy resulted from assisted reproductive technologies, LMP date may be replaced by IUI (intrauterine insemination) or ET (embryo-transfer) date.

* No fetal genetic abnormalities (based on genetic testing, if performed).
* No significant congenital malformations conducted at or beyond 18 weeks of gestation.
* Participants who are willing to provide cord blood.
* Participants who do not plan to give their offspring for adoption or place the child in care.
* Participants who plan to reside in the study area for at least one year after delivery.
* Willing to have their infant followed-up after delivery for a period of 12 months.

Note that women whose pregnancies resulted from Assisted Reproductive Technologies may be enrolled if they meet all inclusion criteria and none of the exclusion criteria.

Infant participants

* Live-born from the study pregnancy.
* If required per local regulations/guidelines, re-signed (confirmed) written or witnessed/thumb printed informed consent for study participation of the infant obtained from the infant's mother and/or father and/or LAR, before performing any study-specific procedure. To comply other protocol required procedures that begin immediately after birth: If written consent cannot be provided by the infant's parent(s)/LAR(s) readily post-birth, verbal consent, if permitted per local regulation, may be sought from the infant's parent(s)/LAR(s) instead. Verbal consent should be documented in the source data by the investigator or delegate. The infant's parent(s)/LAR(s) will provide additional, written informed consent by (or before) Visit 2-NB.

Exclusion Criteria:

Maternal participants

Medical conditions

* History of any reaction or hypersensitivity likely to be exacerbated by any component of the study intervention.
* Hypersensitivity to latex.
* Acute or chronic clinically significant abnormality or poorly controlled pre-existing condition or any other clinical conditions.
* Subjects who have received 2 or more doses of any RSV vaccine in the past.
* Significant complications in the current pregnancy such as:

  * Gestational hypertension at ≥20 weeks of gestation in the absence of proteinuria in a woman with a previously normal blood pressure.
  * Gestational diabetes which is not controlled by medication, diet and/or exercise
  * Pre-eclampsia
  * Eclampsia
  * Intrauterine Growth Restriction/Fetal Growth Restriction
  * Placenta previa
  * Placental abruption, placenta accreta/percreta/increta, chorioamnionitis or any abnormalities
  * Polyhydramnios
  * Oligohydramnios
  * Preterm labor or history of preterm labor in the current pregnancy.
  * Any intervention to prevent preterm delivery or medical treatment for suspected preterm delivery
  * Cholestasis
  * Other pregnancy-related complications
* History of 2 or more prior stillbirths or neonatal deaths, or history of 2 or more preterm births at ≤ 34 weeks gestation, or 3 or more consecutive spontaneous abortions.
* Significant structural abnormalities of the uterus or cervix.
* Known human immunodeficiency virus infection, as assessed by local standard of care serologic tests.
* Known or suspected hepatitis B or C virus infection.
* Known or suspected infection during the current pregnancy with Toxoplasma, Parvovirus B19, Syphilis, Zika, Rubella, Varicella, CMV or primary genital Herpes Simplex.
* Active infection with tuberculosis.
* Any confirmed or suspected immunosuppressive or immunodeficient condition.
* Current autoimmune disorder.
* Lymphoproliferative disorder or malignancy within 5 years before study vaccination.
* Any conditions that, in the investigator's judgement, may interfere with participant's ability to comply with study procedures or receipt of prenatal care.
* Any condition which, in the investigator's opinion, would increase the risks of study participation to the unborn infant.

Prior/Concomitant therapy

* Prior receipt of any RSV vaccine in the current pregnancy or prior receipt of 2 or more doses of any RSV vaccine prior to study vaccination.
* Use of any investigational or non-registered product other than the study vaccine/product, or planned use during the study period).

The exception to this are investigational products administered in the setting of a pandemic.

* Planned administration/administration of any vaccine within 29 days before study vaccine administration (Day -28 to Day 1) or planned administration through delivery, except:

  * Seasonal influenza vaccines, tetanus vaccines, dTpa/Tdap - alone vaccines, dTpa/Tdap vaccines that also contain other antigens and Hepatitis B vaccines, which may be administered ≥ 15 days before or after study vaccination.

    * Note that if public health authorities organize an emergency mass vaccination for an unforeseen public health threat (e.g.: a pandemic) outside the routine immunisation program, then the intervals described above can be reduced if necessary for that mass vaccination vaccine, provided the vaccine is licensed and used according to its Product Information. In that sense, COVID-19 vaccines may be allowed, when administered ≥ 15 days before or after study vaccination.
* Administration of immunoglobulins (except anti-Rh0D IG, which may be administered at any time), blood products or plasma derivatives within 3 months before study vaccination or planned administration through delivery (Visit 3).
* Administration of immune-modifying therapy within 6 months before the study vaccination, or planned administration through delivery.

Prior/Concurrent clinical study experience

* Concurrently participating in another clinical study, at any time during the study period, in which the participant has been or will be exposed to an investigational or a non-investigational intervention.
* Subjects who were lost to follow-up or prematurely withdrawn before Day 43 in the RSV MAT-004, RSV MAT-009 and RSV MAT-012 studies.

Other exclusions

* Alcoholism or substance use disorder within the past 24 months based on the presence of 2 or more abuse criteria.
* A local condition that in the opinion of the Investigator precludes injection of the study vaccine/product or precludes assessment of local (administration site) reactogenicity.
* Consanguinity of maternal participant and her partner.
* Any study personnel or their immediate dependents, family, or household members.

Infant participants

* Concurrently participating in another clinical study, at any time during the study period, in which the participant has been or will be exposed to an investigational or a non-investigational vaccine/product.
* Any condition which, in the investigator's opinion, would increase the risks of study participation to the infant.
* Child in care.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only pregnant women, 18 to 49 YOA are included in the study.
Enrollment: 0 (Actual)
Dates: Start 2022-03-11 (Estimated); Primary Completion 2023-11-06 (Estimated); Study Completion 2024-10-24 (Estimated)

PRIMARY OUTCOMES:
Percentage of maternal participants with solicited administration site events during the 7-day follow-up period after vaccination in the current study | During the 7-day follow-up period after vaccination in the current study (administered at Day 1)
  The following administration site events are solicited for maternal participants: pain, redness and swelling.
Percentage of maternal participants with solicited systemic events during the 7-day follow-up period after vaccination in the current study | During the 7-day follow-up period after vaccination in the current study (administered at Day 1)
  The following systemic events are solicited for maternal participants: fatigue, fever, nausea, vomiting, diarrhea, abdominal pain and headache. Fever is defined as temperature > 38.0°C/100.4°F regardless of the location of measurement. The preferred location for measuring temperature in this study is the oral cavity.
Percentage of maternal participants with unsolicited adverse events (AEs) during the 30-day follow-up period after vaccination in the current study | During the 30-day follow-up period after vaccination in the current study (administered at Day 1)
  Any AE reported in addition to those solicited during the clinical study. Also, any 'solicited' symptom with onset outside the specified period of follow-up for solicited symptoms will be reported as an unsolicited adverse event.
Percentage of maternal participants with serious adverse events (SAEs), AEs leading to study withdrawal and medically attended AEs (MAEs) from Day 1 up to 42 days post-delivery in the current study | From Day 1 up to 42 days post-delivery in the current study
  An SAE is any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study participant or results in abnormal pregnancy outcomes. An MAE is an unsolicited AE for which the participants receive medical attention and is defined as symptoms or illnesses requiring a hospitalization, or an emergency room visit, or visit to/by a health care provider. AE leading to study withdrawal = any AE that leads to withdrawal of the participant from the study.
Percentage of maternal participants with pregnancy outcomes from Day 1 up to 42 days post-delivery in the current study | From Day 1 up to 42 days post-delivery in the current study
  Pregnancy outcomes include live birth with no congenital anomalies, live birth with minor congenital anomalies only, live birth with at least 1 major congenital anomaly, fetal death/still birth (antepartum or intrapartum) with no congenital anomalies, fetal death/still birth (antepartum or intrapartum) with only minor congenital anomalies, fetal death/still birth (antepartum or intrapartum) with at least 1 major congenital anomaly, elective/therapeutic termination with no congenital anomalies, elective/therapeutic termination with only minor congenital anomalies and elective/therapeutic termination with at least 1 major congenital anomaly.
Percentage of maternal participants with pregnancy-related adverse events of special interest (AESIs) from Day 1 up to 42 days post-delivery in the current study | From Day 1 up to 42 days post-delivery in the current study
  Pregnancy-related AESIs include maternal death, hypertensive disorders of pregnancy (gestational hypertension, pre-eclampsia, pre-eclampsia with severe features including eclampsia), fetal growth restriction, gestational diabetes mellitus, pathways to preterm birth (premature preterm rupture of membranes, preterm labor, provider-initiated preterm birth) and chorioamnionitis.
Percentage of infant participants with neonatal / infant AESIs from birth up to 42 days post-birth in the current study | From birth up to 42 days post-birth in the current study
  Neonatal / infant AESIs include small for gestational age, low birth weight including very low and extremely low birth weight, congenital anomalies, neonatal death and preterm birth.
Percentage of infant participants with SAEs, (S)AEs leading to study withdrawal and MAEs from birth up to 42 days post-birth in the current study | From birth up to 42 days post-birth in the current study
  An SAE is any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study participant or results in abnormal pregnancy outcomes. An MAE is an unsolicited AE for which the participants receive medical attention and is defined as symptoms or illnesses requiring a hospitalization, or an emergency room visit, or visit to/by a health care provider. (S)AE leading to study withdrawal = any (S)AE that leads to withdrawal of the participant from the study.
RSV MAT immunoglobulin G (IgG)-specific antibody geometric mean concentrations (GMCs) for maternal participants at Day 31 post-vaccination in the current study | At Day 31 post-vaccination in the current study
  IgG antibody concentrations against RSV MAT are measured by enzyme-linked immunosorbent assay (ELISA). This outcome measure is evaluated between participants enrolled in Prior_RSV MAT group and Prior_Placebo group.
RSV MAT IgG-specific antibody GMCs for maternal participants at delivery in the current study | At delivery in the current study
  IgG antibody concentrations against RSV MAT are measured by ELISA. This outcome measure is evaluated between participants enrolled in Prior_RSV MAT group and Prior_Placebo group.
RSV-A neutralizing antibody geometric mean titers (GMTs) for maternal participants at Day 31 post-vaccination in the current study | At Day 31 post-vaccination in the current study
  Serum antibody titers against RSV-A are measured by neutralization assay. This outcome measure is evaluated between participants enrolled in Prior_RSV MAT group and Prior_Placebo group.
RSV-A neutralizing antibody GMTs for maternal participants at delivery in the current study | At delivery in the current study
  Serum antibody titers against RSV-A are measured by neutralization assay. This outcome measure is evaluated between participants enrolled in Prior_RSV MAT group and Prior_Placebo group.
RSV-B neutralizing antibody GMTs for maternal participants at Day 31 post-vaccination in the current study | At Day 31 post-vaccination in the current study
  Serum antibody titers against RSV-B are measured by neutralization assay. This outcome measure is evaluated between participants enrolled in Prior_RSV MAT group and Prior_Placebo group.
RSV-B neutralizing antibody GMTs for maternal participants at delivery in the current study | At delivery in the current study
  Serum antibody titers against RSV-B are measured by neutralization assay. This outcome measure is evaluated between participants enrolled in Prior_RSV MAT group and Prior_Placebo group.

SECONDARY OUTCOMES:
Percentage of maternal participants with SAEs and AEs leading to study withdrawal from Day 1 up to Day 181 post-delivery in the current study | From Day 1 up to Day 181 post-delivery in the current study
  An SAE is any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study participant or results in abnormal pregnancy outcomes. AE leading to study withdrawal = any AE that leads to withdrawal of the participant from the study.
Percentage of maternal participants in Prior_RSV MAT group with solicited administration site events during the 7-day follow-up period after administration of the first and repeat vaccination | During the 7-day follow-up period after administration of the first vaccination (administered at Day 1 in NCT04126213, NCT04605159 or NCT04980391 studies) and the repeat vaccination (administered at Day 1 in the current study)
  The following administration site events are solicited for maternal participants: pain, redness and swelling.
Percentage of maternal participants in Prior_RSV MAT group with solicited systemic events during the 7-day follow-up period after administration of the first and repeat vaccination | During the 7-day follow-up period after administration of the first vaccination (administered at Day 1 in NCT04126213, NCT04605159 or NCT04980391 studies) and repeat vaccination (administered at Day 1 in the current study)
  The following systemic events are solicited for maternal participants: fatigue, fever, nausea, vomiting, diarrhea, abdominal pain and headache. Fever is defined as temperature > 38.0°C/100.4°F regardless of the location of measurement. The preferred location for measuring temperature in this study is the oral cavity.
Percentage of maternal participants in Prior_RSV MAT group with unsolicited AEs during the 30-day follow-up period after administration of the first and repeat vaccination | During the 30-day follow-up period after administration of the first vaccination (administered at Day 1 in NCT04126213, NCT04605159 or NCT04980391 studies) and repeat vaccination (administered at Day 1 in the current study)
  Any AE reported in addition to those solicited during the clinical study. Also, any 'solicited' symptom with onset outside the specified period of follow-up for solicited symptoms will be reported as an unsolicited adverse event.
Percentage of maternal participants in Prior_RSV MAT group with SAEs and AEs leading to study withdrawal from Day 1 up to Day 181 post-delivery after administration of the first and repeat vaccination | From Day 1 up to Day 181 post-delivery after administration of the first vaccination in NCT04126213, NCT04605159 or NCT04980391 studies and repeat vaccination in the current study
  An SAE is any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study participant or results in abnormal pregnancy outcomes. AE leading to study withdrawal = any AE that leads to withdrawal of the participant from the study.
Percentage of maternal participants in Prior_RSV MAT group with MAEs from Day 1 up to 42 days post-delivery after administration of the first and the repeat vaccination | From Day 1 up to 42 days post-delivery after administration of the first vaccination in NCT04126213, NCT04605159 or NCT04980391 studies and repeat vaccination in the current study
  An MAE is an unsolicited AE for which the participants receive medical attention and is defined as symptoms or illnesses requiring a hospitalization, or an emergency room visit, or visit to/by a health care provider.
Percentage of maternal participants in Prior_RSV MAT group with pregnancy outcomes from Day 1 up to 42 days post-delivery after administration of the first and repeat vaccination | From Day 1 up to 42 days post-delivery after administration of the first vaccination in NCT04126213, NCT04605159 or NCT04980391 studies and repeat vaccination in the current study
  Pregnancy outcomes include live birth with no congenital anomalies, live birth with minor congenital anomalies only, live birth with at least 1 major congenital anomaly, fetal death/still birth (antepartum or intrapartum) with no congenital anomalies, fetal death/still birth (antepartum or intrapartum) with only minor congenital anomalies, fetal death/still birth (antepartum or intrapartum) with at least 1 major congenital anomaly, elective/therapeutic termination with no congenital anomalies, elective/therapeutic termination with only minor congenital anomalies and elective/therapeutic termination with at least 1 major congenital anomaly.
Percentage of maternal participants in Prior_RSV MAT group with pregnancy-related AESIs from Day 1 up to 42 days post-delivery after administration of the first and repeat vaccination | From Day 1 up to 42 days post-delivery after administration of the first vaccination in NCT04126213, NCT04605159 or NCT04980391 studies and repeat vaccination in the current study
  Pregnancy-related AESIs include maternal death, hypertensive disorders of pregnancy (gestational hypertension, pre-eclampsia, pre-eclampsia with severe features including eclampsia), fetal growth restriction, gestational diabetes mellitus, pathways to preterm birth (premature preterm rupture of membranes, preterm labor, provider-initiated preterm birth) and chorioamnionitis.
Percentage of infant participants with SAEs, (S)AEs leading to study withdrawal and MAEs from birth up to Day 366 post-birth in the current study | From birth up to Day 366 post-birth in the current study
  An SAE is any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study participant or results in abnormal pregnancy outcomes. An MAE is an unsolicited AE for which the participants receive medical attention and is defined as symptoms or illnesses requiring a hospitalization, or an emergency room visit, or visit to/by a health care provider. (S)AE leading to study withdrawal = any (S)AE that leads to withdrawal of the participant from the study.
RSV MAT IgG-specific antibody GMCs for maternal participants in Prior_RSV MAT group at Day 31 post-repeat and first vaccination | At Day 31 post-repeat vaccination administered in the current study and first vaccination administered in NCT04126213, NCT04605159 or NCT04980391 studies
  This outcome measure is evaluated within the participants enrolled in Prior_RSV MAT group.
RSV MAT IgG-specific antibody GMCs for maternal participants in Prior_RSV MAT group at delivery post-repeat and first vaccination | At delivery post-repeat vaccination administered in the current study and first vaccination administered in NCT04126213, NCT04605159 or NCT04980391 studies
  This outcome measure is evaluated within the participants enrolled in Prior_RSV MAT group.
RSV-A neutralizing antibody GMTs for maternal participants in Prior_RSV MAT group at Day 31 post-repeat and first vaccination | At Day 31 post-repeat vaccination administered in the current study and first vaccination administered in NCT04126213, NCT04605159 or NCT04980391 studies
  This outcome measure is evaluated within the participants enrolled in Prior_RSV MAT group.
RSV-A neutralizing antibody GMTs for maternal participants in Prior_RSV MAT group at delivery post-repeat and first vaccination | At delivery post-repeat vaccination administered in the current study and first vaccination administered in NCT04126213, NCT04605159 or NCT04980391 studies
  This outcome measure is evaluated within the participants enrolled in Prior_RSV MAT group.
RSV-B neutralizing antibody GMTs for maternal participants in Prior_RSV MAT group at Day 31 post-repeat and first vaccination | At Day 31 post-repeat vaccination administered in the current study and first vaccination administered in NCT04126213, NCT04605159 or NCT04980391 studies
  This outcome measure is evaluated within the participants enrolled in Prior_RSV MAT group.
RSV-B neutralizing antibody GMTs for maternal participants in Prior_RSV MAT group at delivery post-repeat and first vaccination | At delivery post-repeat vaccination administered in the current study and first vaccination administered in NCT04126213, NCT04605159 or NCT04980391 studies
  This outcome measure is evaluated within the participants enrolled in Prior_RSV MAT group.
Geometric mean ratio between cord blood and maternal RSV MAT IgG-specific antibody concentrations at delivery in the current study | At delivery in the current study
  Transfer of RSV-specific antibodies from maternal participants vaccinated with the RSV MAT vaccine to their infants is calculated as the ratio between cord blood and maternal RSV MAT IgG-specific antibody concentrations. Cord blood or infant blood sample is collected within 3 days after birth (if no cord blood sample can be obtained).
RSV MAT IgG-specific antibody GMCs for infant participants at delivery in the current study | At delivery in the current study
  IgG antibody concentrations against RSV MAT are measured by ELISA.
RSV-A neutralizing antibody GMTs for infant participants at delivery in the current study | At delivery in the current study
  Serum antibody titers against RSV-A are measured by neutralization assay.
RSV-B neutralizing antibody GMTs for infant participants at delivery in the current study | At delivery in the current study
  Serum antibody titers against RSV-B are measured by neutralization assay.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- United States (2):
  - GSK Investigational Site, Missoula, Montana
  - GSK Investigational Site, Norfolk, Nebraska

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, a key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.